CLINICAL TRIAL: NCT02931253
Title: Metformin as an Upstream Therapy in Atrial Fibrillation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issue: Enrollment expectation not met
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1602-01
Record Dates: First submitted 2016-10-07; First posted 2016-10-13 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin Group (Experimental): Metformin 500 mg daily initiated 6 weeks prior to scheduled ablation.
  Metformin increased to 2000 mg daily (1000 mg twice a day) as tolerated over the initial 3 weeks.
  Interventions: Drug: Metformin
- Control Group (No Intervention): Standard of care - ablation only

INTERVENTIONS:
Drug: Metformin — Metformin will be started as one pill (500 mg metformin) once a day with a meal. If the subject has no side effects from this dose, the dose will be increased to two pills (1000 mg) twice a day to be taken with meals.
  Arms: Metformin Group

SUMMARY:
The purpose of this study is to see if the study drug metformin will help patients who are overweight and have atrial fibrillation. This study aims to see if metformin helps patients stay in normal sinus rhythm after a catheter ablation.

Metformin is investigational for use in patients with atrial fibrillation. Metformin is approved by the Food and Drug Administration (FDA) for use in patients with type 2 Diabetes Mellitus. Metformin is used with a proper diet and exercise program to control high blood sugar, and has been shown to help people lose weight. This study aims to look at the effects of metformin on weight loss and heart rhythm in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Enrollment: Consent, medical history, and dietary education. Randomization. treatment Metformin 500mg daily and increased as tolerated to 2000 mg daily over three weeks or control -no treatment. 6 weeks. Pre procedure safety labs, EKG, Atrial Fibrillation Severity Score survey, metformin held 48 hours prior to rhythm control procedure. Treatment resumed 48 hours post procedure or when renal function at baseline. Treatment plan for 6 months or discontinuation at any time they are found to meet the baseline exclusion criteria. Follow-up at 3 month and 6 month post procedure. Continuation of treatment at study completion determined by primary cardiologist or care provider.

ELIGIBILITY:
Inclusion Criteria:

* All individuals diagnosed with Atrial Fibrillation and choosing to undergo a rhythm control strategy at Robert Packer Hospital with a BMI ≥ 27 will be eligible for the study. All subjects must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Individuals who are already taking metformin or other antidiabetic medications including insulin, have a diagnosis of diabetes, have a known allergy or FDA-labeled contraindication to taking metformin, eGFR below 30 mL/min per 1.73 m2 or other clinical diagnosis of advanced renal disease,, have acute or chronic metabolic acidosis (serum bicarbonate <22 mEq/L), have a history of significant alcohol use (>2 drinks/day on average), have a history of hepatic dysfunction (serum bilirubin 1.5X greater than the upper limit of normal), have a history of New York Heart Association (NYHA) Class III or IV heart failure, or are pregnant will be excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Guthrie Clinic, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated prior to meeting enrollment target. Enrollment rate slower than expected.
Groups:
- Metformin Group: Metformin 500 mg daily initiated 6 weeks prior to scheduled ablation.
  Metformin increased to 2000 mg daily (1000 mg twice a day) as tolerated over the initial 3 weeks.
  Metformin: Metformin will be started as one pill (500 mg metformin) once a day with a meal. If the subject has no side effects from this dose, the dose will be increased to two pills (1000 mg) twice a day to be taken with meals.
Period: Overall Study
Arm/Group | Metformin Group | Control Group
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Group | Control Group | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (4) | 65 (3) | 66 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Maintain Sinus Rhythm
Description: Number of participants who maintain sinus rhythm, normal heart rhythm by electrocardiogram (ECG)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
Participants | 1 | 0

2. Secondary Outcome: Number of Participants Requiring Hospitalization
Description: Hospitalization related to arrhythmic events or medication side effects
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Requiring Antiarrhythmic Medications
Description: Total count of participants on anti-arrhythmic medications
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
Participants | 1 | 1

4. Secondary Outcome: Number of Participants Requiring Repeat Ablations
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

5. Secondary Outcome: Change in BMI
Description: Average change in BMI from baseline to 6 month.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
kg/m^2 | 1.8 (.8) | 1.7 (1.3)

6. Secondary Outcome: Hemoglobin A1c
Description: Change from baseline to 6 month
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
percent glycosylated hemoglobin | .1 (.14) | .15 (.1)

7. Secondary Outcome: Number of Participants With Thromboembolic Events
Description: Number of participants who have a thromboembolic event from baseline to 6 months
Time Frame: from baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

8. Other Pre Specified Outcome: Weight Loss
Description: Weight change from baseline to 6 months.
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Metformin Group | Control Group
Number analyzed (Participants) | 2 | 4
pounds | 2 (6.3) | -.6 (3.4)

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | Metformin Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT02931253/Prot_SAP_000.pdf